CLINICAL TRIAL: NCT04402372
Title: Comparative Clinical Efficacy of Novel Bidirectional Peripheral Artery Cannula in Minimally Invasive Aortic Valve Surgery
Brief Title: Novel Bidirectional Peripheral Artery Cannula in Minimally Invasive Aortic Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Serdar Günaydın, Professor, Ankara City Hospital Bilkent
Other Study IDs: 2020-1994
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Efficacy and Safety of Novel Bidirectional Cannula
Keywords: cannula; cardiopulmonary bypass; bidirectional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 30 patients undergoing aortic valve replacement with minimally invasive technique prospectively randomized to receive 19 F bidirectional (BiflowTM, LivaNova, Italy) for femoral artery cannulation
  Interventions: Device: Novel bidirectional cannula (BiflowTM, LivaNova, Italy)
- Group 2: 30 patients undergoing aortic valve replacement with minimally invasive technique prospectively randomized to receive 19 F conventional (HLS, Maquet, Germany cannula with downstream line (6F) for femoral artery cannulation
  Interventions: Device: Novel bidirectional cannula (BiflowTM, LivaNova, Italy)

INTERVENTIONS:
Device: Novel bidirectional cannula (BiflowTM, LivaNova, Italy) — We are going to evaluate the safety and efficacy of the novel bidirectional cannula (BiflowTM, LivaNova, Italy) with specific design to ensure stable distal perfusion compared to conventional cannula with downstream line in patients undergoing femoral arterial cannulation for CPB during minimally invasive surgery

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of the novel bidirectional cannula (BiflowTM, LivaNova, Italy) with specific design to ensure stable distal perfusion compared to conventional cannula with downstream line in patients undergoing femoral arterial cannulation for cardiopulmonary bypass during minimally invasive surgery

DETAILED DESCRIPTION:
The femoral artery is a common site for peripheral cannulation in patients requiring cardiopulmonary bypass (CPB) for minimally invasive cardiac surgical procedures (MICS), redo cardiac surgical procedures, and procedures involving the thoracic aorta Limb ischemia is the most common acute and late vascular complication and has been reported in 10% to 70% of patients Traditional methods to maintain distal perfusion include the use of a downstream cannula or sewing on a side graft, but these techniques are cumbersome, time-consuming, and require additional equipment As a result, current practice is relying on the very small volume of blood that will flow around the cannula and collateral circulation to keep the leg viable, but by the time ischemia is clinically evident, irreversible cell damage may have already occurred The aim of this study is to evaluate the safety and efficacy of the novel bidirectional cannula (BiflowTM, LivaNova, Italy) with specific design to ensure stable distal perfusion compared to conventional cannula with downstream line in patients undergoing femoral arterial cannulation for CPB during MICS

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing minimally invasvie aortic valve replacement 50-90 years of age

Exclusion Criteria:

* previous vascular surgery of the femoral artery, emergency cardiac surgery including type A aortic dissections, internal diameter of the common femoral artery less than 7.5 mm and where the clinician felt adequate flow rates and line pressures would not be achievable with a 19F cannula, because of the patient's weight and body surface area

Ages: 50 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective minimally invasive aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Vascular complications | one moth
  infection, emboli, hematoma, bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Gunaydin, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marasco SF, Tutungi E, Vallance SA, Udy AA, Negri JC, Zimmet AD, McGiffin DC, Pellegrino VA, Moshinsky RA. A Phase 1 Study of a Novel Bidirectional Perfusion Cannula in Patients Undergoing Femoral Cannulation for Cardiac Surgery. Innovations (Phila). 2018 Mar/Apr;13(2):97-103. doi: 10.1097/IMI.0000000000000489. PMID 29697598